CLINICAL TRIAL: NCT06166446
Title: Comparison of Denture Base Adaptation and Per-implant Tissue Health Between CAD and CAM Implant Retained Complete Overdenture
Brief Title: Comparison of Denture Base Adaptation and Per-iimplant Tissue Health Between CAD and CAM Implant Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: A10080921
Record Dates: First submitted 2023-12-03; First posted 2023-12-12 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-11

CONDITIONS: Periimplantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Subtractive Hybridization Techniques

STUDY DESIGN:
Intervention Model Description: 15 completely edentulous patients, divided into two groups, received two implants in the mandibular canine area with ball attachment. The first group received a CAD/CAM-milled mandibular overdenture and a maxillary acrylic conventional complete denture, while the second group received a 3D-printed mandibular overdenture and a maxillary acrylic complete denture. Peri-implant soft tissue was evaluated using clinical parameters including the gingival index, plaque index, bleeding index, and probing depth at the time of mandibular complete overdenture insertion (T0), six months (T6), and twelve months (T12) of denture use.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a CAD/CAM-milled mandibular overdenture and a maxillary acrylic conventional complete denture (Active Comparator): patients received lower denture fabricated by milling technique
  Interventions: Device: subtractive technique
- 3rd printed mandibular overdenture and a maxillary acrylic conventional complete denture (Active Comparator): The denture base was fabricated by adding the material layer by layer
  Interventions: Device: additive technique

INTERVENTIONS:
Device: subtractive technique — The milled denture teeth are then bonded into the milled recesses using a special PMMA bonding system.
  Arms: a CAD/CAM-milled mandibular overdenture and a maxillary acrylic conventional complete denture
Device: additive technique — The denture teeth were printed as one unit using the same method with tooth resin (DENTCA Denture Tooth, Shade A2).
  Arms: 3rd printed mandibular overdenture and a maxillary acrylic conventional complete denture

SUMMARY:
Background: Complete overdenture manufacturing has been greatly developed using computer-aided designing and computer-aided manufacturing (CAD-CAM) technology.

Material and method: 15 completely edentulous patients, divided into two groups, received two implants in the mandibular canine area with ball attachment. The first group received a CAD/CAM-milled mandibular overdenture and a maxillary acrylic conventional complete denture, while the second group received a 3D-printed mandibular overdenture and a maxillary acrylic complete denture. Peri-implant soft tissue and denture adaptation were evaluated using clinical parameters

DETAILED DESCRIPTION:
Background: In recent years, complete overdenture manufacturing has been greatly developed using computer-aided designing and computer-aided manufacturing (CAD-CAM) technology. This clinical study compared the soft tissue health between CAD/CAM-milled and 3D-printed implants that retained complete overdentures.

Material and method: 15 completely edentulous patients, divided into two groups, received two implants in the mandibular canine area with ball attachment. The first group received a CAD/CAM-milled mandibular overdenture and a maxillary acrylic conventional complete denture, while the second group received a 3D-printed mandibular overdenture and a maxillary acrylic complete denture. Peri-implant soft tissue was evaluated using clinical parameters including the gingival index, plaque index, bleeding index, and probing depth at the time of mandibular complete overdenture insertion (T0), six months (T6), and twelve months (T12) of denture use.

ELIGIBILITY:
Inclusion Criteria:

poor denture adaptation co-operative patients

Exclusion Criteria:

metabolic diseases uncontrolled diabetes osteoporosis and hyperparathyroidism.

Ages: 58 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Modified Plaque Index | 12 months
  a calibrated pressure sensitive plastic periodontal probe, the distance between marginal border of the peri-implant mucosa and the tip of the probe was measured and considered as pocket depth

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Aboelez, Phd, Principal Investigator — Mansoura University; Radwa Emera, Phd, Study Director — Mansoura University
Locations (1):
- Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Emera RMK, Shady M, Alnajih MA. Comparison of retention and denture base adaptation between conventional and 3D-printed complete dentures. J Dent Res Dent Clin Dent Prospects. 2022 Summer;16(3):179-185. doi: 10.34172/joddd.2022.030. Epub 2022 Nov 15. PMID 36704186